CLINICAL TRIAL: NCT06494111
Title: Systemic Therapy of Open-label Prophylactic Pravastatin or Pentoxifylline/Tocopherol Prevention of Lymphedema Advancing to Eventual Fibrosis: an Interventional Registry-embedded Bayesian Randomized Trial for Radiation Sequelae (STOP4-LATE-FIBROSE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0968; NCI-2024-05763 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema; Fibrosis
MeSH Terms: conditions — Lymphedema; Fibrosis | interventions — Pravastatin; Pentoxifylline; Tocopherols; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Beginning at 6 months after radiation therapy, participants will take 40 mg pravastatin by mouth 1 time a day for about 12 months.
  Interventions: Drug: Pravastatin
- Group 2 (Experimental): Beginning at 6 months after radiation therapy, participants will take pentoxifylline and vitamin E by mouth 3 times a day for about 12 months.
  Interventions: Drug: Pentoxifylline; Drug: Tocopherol
- Group 3 (No Intervention): Participants will not be given any of the study drugs, as this is the control group.

INTERVENTIONS:
Drug: Pravastatin — Given by PO
  Arms: Group 1
Drug: Pentoxifylline — Given by PO
  Arms: Group 2
Drug: Tocopherol — Given by PO
  Other Names: Vitamin E
  Arms: Group 2

SUMMARY:
To learn if pentoxifylline and vitamin E or pravastatin can reduce radiation-induced lymphedema/fibrosis.

DETAILED DESCRIPTION:
* Primary Objectives Determine the relative utility of pentoxifylline/tocopherol or pravastatin to reduce clinician-rated radiation lymphedema/fibrosis.
* Secondary Objectives Determine the relative effect size observed of pentoxifylline/tocopherol or pravastatin to reduce objective imaging-derived measures of radiation lymphedema/fibrosis-related sequalae.

Determine the relative effect size observed of pentoxifylline/tocopherol or pravastatin to reduce patient-reported measures of toxicity associated with lymphedema/fibrosis-related sequalae.

ELIGIBILITY:
Inclusion Criteria:

• Untreated T0-T4N0-3M0 oropharyngeal squamous carcinoma.

1. Dispositioned to radiotherapy with prescribed dose to unilateral or bilateral neck(s).
2. Creatinine clearance >30mL/min
3. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of pentoxifylline/pravastatin in participants <18 years of age, children are excluded from this study
4. ECOG performance status ≤2 (Karnofsky ≥60%,)
5. Participants must have adequate organ and marrow function as defined below

   * absolute neutrophil count ≥1,000/mcL
   * platelets ≥100,000/mcL
   * total bilirubin ≤ institutional upper limit of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤3 x institutional ULN
   * creatinine ≤1.5 x institutional ULN
6. The effects of pentoxifylline/pravastatin on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following.

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.
   * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Active liver disease (Child-Pugh class B-C), cirrhosis, nor active alcoholism.
2. History of myopathy/rhabdomyolysis.
3. History of acute myocardial infarction or severe coronary disease.
4. Pregnant/post-menopausal, or male.
5. History of diabetes mellitus.
6. Allergy/hypersensitivity to Hydroxymethylglutaryl-coenzyme A (HMG Co-A) reductase inhibitor and/or xanthine derivatives, e.g., caffeine, theophylline, theobromine.
7. Contraindications for MRI
8. Participants who are receiving any other investigational agents.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to statins, hemorheologic agents or other agents used in study
10. Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Fuller, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org